CLINICAL TRIAL: NCT05217667
Title: Phase 2 Study to Evaluate the Safety and Efficacy of ARO-ANG3 in Subjects With Homozygous Familial Hypercholesterolemia (HOFH)
Brief Title: Study of ARO-ANG3 in Participants With Homozygous Familial Hypercholesterolemia (HOFH)
Acronym: Gateway
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Arrowhead Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AROANG3-2003
Record Dates: First submitted 2022-01-20; First posted 2022-02-01 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Homozygous Familial Hypercholesterolemia
MeSH Terms: conditions — Homozygous Familial Hypercholesterolemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ARO-ANG3 Dose 1 (Experimental): ARO-ANG3 Dose Level 1 subcutaneous (SC)
  Interventions: Drug: ARO-ANG 3 Injection
- ARO-ANG3 Dose 2 (Experimental): ARO-ANG3 Dose Level 2 SC
  Interventions: Drug: ARO-ANG 3 Injection

INTERVENTIONS:
Drug: ARO-ANG 3 Injection — Participants will be randomized to receive ARO-ANG3 SC on Day 1 and Day 84 during the initial 36 Weeks of the study and on Day1 and Months 3, 6, 9, 12, 15, 18, and 21 of the extension period

SUMMARY:
Participants with documented homozygous familial hypercholesterolemia (HoFH) who have provided informed consent will receive 2 open-label doses of ARO-ANG3 and be evaluated for safety and efficacy parameters through 36 weeks. Participants who complete the first 36 week treatment period may opt to continue in an additional 24-month extension period during which they will receive up to 8 doses open-label doses of ARO-ANG3.

ELIGIBILITY:
Inclusion Criteria:

* Fasting LDL-C >100 mg/dL at Screening
* Weight of ≥ 40 kg and body mass index ≥ 18.5 and ≤ 40 kg/m2
* Diagnosis of HoFH based on a supportive genetic test or clinical diagnosis
* On stable maximally tolerated lipid lowering therapy
* Willing to abide by stable low-fat, low-cholesterol, heart-healthy diet for at least 4 weeks prior to Day 1
* Participants of childbearing potential (males & females) must agree to use highly-effective contraception during the study and for at least 24 weeks from the last dose of study medication.
* Women of childbearing potential must have a negative pregnancy test and cannot be breastfeeding
* Women of childbearing potential on hormonal contraceptives must be stable on the medications for > 2 menstrual cycles prior to Day 1
* Willing to provide written informed consent and to comply with study requirements

Exclusion Criteria:

* Current use or use within 365 days from Day 1 of any hepatocyte targeted small interfering RNA oligonucleotides (siRNA) or antisense oligonucleoside molecule
* Use of evinacumab (some exceptions apply)
* Fasting TG > 300 mg/dL at Screening
* Presence of any clinically significant uncontrolled endocrine disease known to influence serum lipids or lipoproteins
* Newly diagnosed (within 3 months prior to informed consent) or poorly controlled diabetes (Hemoglobin A1c > 9%)
* Use of systemic corticosteroids (some exceptions apply)
* Symptoms of myocardial ischemia or severe left ventricular dysfunction
* History of metastatic malignancy within 3 years of Day 1 (some exceptions apply)
* Planned cardiac procedure/surgery such as coronary artery bypass graft (CABG) surgery, percutaneous coronary intervention (PCI), carotid surgery or stenting, or carotid revascularization

Note: additional inclusion/exclusion criteria may apply per protocol

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Percent Change from Baseline in Fasting Calculated Low-Density Lipoprotein-Cholesterol (LDL-C) and LDL-C by Preparative Ultracentrifugation (LDL-C [PUC]) up to Week 24 | Baseline, up to Week 24

SECONDARY OUTCOMES:
Percent Change from Baseline in Fasting LDL-C (PUC) Over Time | Baseline, up to Week 36 (initial treatment period), up to Month 24 (extension period)
Absolute Change from Baseline in Fasting LDL-C (PUC) Over Time | Baseline, up to Week 36 (initial treatment period), up to Month 24 (extension period)
Percent Change from Baseline in Fasting Calculated LDL-C Over Time | Baseline, up to Week 36 (initial treatment period), up to Month 24 (extension period)
Absolute Change from Baseline in Fasting Calculated LDL-C Over Time | Baseline, up to Week 36 (initial treatment period), up to Month 24 (extension period)
Percent Change from Baseline in Fasting Angiopoietin-like 3 (ANGPTL3) Over Time | Baseline, up to Week 36 (initial treatment period), up to Month 24 (extension period)
Absolute Change from Baseline in Fasting ANGPTL3 Over Time | Baseline, up to Week 36 (initial treatment period), up to Month 24 (extension period)
Percent Change from Baseline in Fasting Total Apolipoprotein B (ApoB) Over Time | Baseline, up to Week 36 (initial treatment period), up to Month 24 (extension period)
Absolute Change from Baseline in Fasting Total ApoB Over Time | Baseline, up to Week 36 (initial treatment period), up to Month 24 (extension period)
Percent Change from Baseline in Fasting High-Density Lipoprotein-Cholesterol (HDL-C) Over Time | Baseline, up to Week 36 (initial treatment period), up to Month 24 (extension period) 36
Absolute Change from Baseline in Fasting HDL-C Over Time | Baseline, up to Week 36 (initial treatment period), up to Month 24 (extension period)
Percent Change from Baseline in Fasting Non-High-Density Lipoprotein-Cholesterol (Non-HDL-C) Over Time | Baseline, up to Week 36 (initial treatment period), up to Month 24 (extension period)
Absolute Change from Baseline in Fasting Non-HDL-C Over Time | Baseline, up to Week 36 (initial treatment period), up to Month 24 (extension period)
Percent Change from Baseline in Fasting Very-Low-Density Lipoprotein-Cholesterol (VLDL-C) Over Time | Baseline, up to Week 36 (initial treatment period), up to Month 24 (extension period)
Absolute Change from Baseline in VLDL-C Over Time | Baseline, up to Week 36 (initial treatment period), up to Month 24 (extension period)
Percent Change from Baseline in Fasting Total Cholesterol (TC) Over Time | Baseline, up to Week 36 (initial treatment period), up to Month 24 (extension period)
Absolute Change from Baseline in Fasting TC Over Time | Baseline, up to Week 36 (initial treatment period), up to Month 24 (extension period)
Percent Change from Baseline in Fasting Triglycerides (TG) Over Time | Baseline, up to Week 36 (initial treatment period), up to Month 24 (extension period)
Absolute Change from Baseline in Fasting TG Over Time | Baseline, up to Week 36 (initial treatment period), up to Month 24 (extension period)
Number of Participants with Treatment Emergent Adverse Events (TEAEs) | Baseline, up to Week 36 (initial treatment period), up to Month 24 (extension period)
Number of Participants with Anti-Drug Antibodies (ADAs) to ARO-ANG3 Over Time | Baseline, up to Week 36 (initial treatment period), up to Month 24 (extension period)
Proportion of Participants meeting United States National Lipid Association Apheresis Eligibility Criteria of LDL-C ≥ 300 mg/dL at Week 24 | Week 24
Proportion of Participants Meeting European Union (EU) Apheresis Eligibility Criteria per German Apheresis Working Group at Week 24 | Week 24

CONTACTS AND LOCATIONS:
Locations (7):
- United States (2):
  - Research Site 4, Mount Sinai, New York
  - Research Site 5, Cincinnati, Ohio
- Australia (2):
  - Research Site 8, Camperdown, New South Wales
  - Research Site 3, Nedlands, Western Australia
- Canada (2):
  - Research Site 2, Chicoutimi, Quebec
  - Research Site 1, Québec, Quebec
- Research Site 7, Johannesburg, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Raal FJ, Bergeron J, Gaudet D, Rosenson RS, Sullivan DR, Turner T, Hegele RA, Ballantyne CM, Knowles JW, Leeper NJ, Goldberg IJ, Zhou R, Muhsin M, Hellawell J, Hamilton J, Watts GF. Zodasiran, an RNAi therapeutic targeting ANGPTL3, for treating patients with homozygous familial hypercholesterolaemia (GATEWAY): an open-label, randomised, phase 2 trial. Lancet Diabetes Endocrinol. 2026 Feb;14(2):123-136. doi: 10.1016/S2213-8587(25)00290-6. Epub 2025 Dec 18. PMID 41422812
- [Derived] Dimitriadis K, Theofilis P, Iliakis P, Pyrpyris N, Dri E, Sakalidis A, Soulaidopoulos S, Tsioufis P, Fragkoulis C, Chrysohoou C, Tsiachris D, Tsioufis K. Management of dyslipidemia in coronary artery disease: the present and the future. Coron Artery Dis. 2024 Sep 1;35(6):516-524. doi: 10.1097/MCA.0000000000001375. Epub 2024 Apr 29. PMID 38682459